CLINICAL TRIAL: NCT04480736
Title: A Phase 2a, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Antiviral Activity, Safety, and Pharmacokinetics of Repeated Oral Doses of JNJ-64281802 Against Dengue Serotype 1 Infection in a Dengue Human Challenge Model in Healthy Adult Participants
Brief Title: A Study of JNJ-64281802 Against Dengue Serotype 1 Infection in a Dengue Human Challenge Model in Healthy Adult Participants
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: portfolio reprioritization
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CR108700; 64281802DNG2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-07-17; First posted 2020-07-21 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Placebo (Placebo Comparator): Participants will receive matching placebo of JNJ-64281802 orally.
  Interventions: Drug: Placebo
- JNJ-64281802 High dose (Experimental): Participants will receive high dose of JNJ-64281802 orally.
  Interventions: Drug: JNJ-64281802 High dose
- JNJ-64281802 Medium dose (Experimental): Participants will receive medium dose of JNJ-64281802 orally.
  Interventions: Drug: JNJ-64281802 Medium dose
- JNJ-64281802 Low dose (Experimental): Participants will receive low dose of JNJ-64281802 orally.
  Interventions: Drug: JNJ-64281802 Low dose
- JNJ-64281802 Dosing Regimen X (Experimental): Participants will receive dosing regimen X of JNJ-64281802 orally.
  Interventions: Drug: JNJ-64281802 Dosing Regimen X
- JNJ-64281802 Dosing Regimen Y (Experimental): Participants will receive dosing regimen Y of JNJ-64281802 orally.
  Interventions: Drug: JNJ-64281802 Dosing Regimen Y
- JNJ-64281802 Dosing Regimen Z (Experimental): Participants will receive dosing regimen Z of JNJ-64281802 orally.
  Interventions: Drug: JNJ-64281802 Dosing Regimen Z

INTERVENTIONS:
Drug: Placebo — Matching placebo will be administered orally.
  Arms: Placebo
Drug: JNJ-64281802 High dose — JNJ-64281802 high dose will be administered orally.
  Arms: JNJ-64281802 High dose
Drug: JNJ-64281802 Medium dose — JNJ-64281802 medium dose will be administered orally.
  Arms: JNJ-64281802 Medium dose
Drug: JNJ-64281802 Low dose — JNJ-64281802 low dose will be administered orally.
  Arms: JNJ-64281802 Low dose
Drug: JNJ-64281802 Dosing Regimen X — JNJ-64281802 dosing regimen X will be administered orally.
  Arms: JNJ-64281802 Dosing Regimen X
Drug: JNJ-64281802 Dosing Regimen Y — JNJ-64281802 dosing regimen Y will be administered orally.
  Arms: JNJ-64281802 Dosing Regimen Y
Drug: JNJ-64281802 Dosing Regimen Z — JNJ-64281802 dosing regimen Z will be administered orally.
  Arms: JNJ-64281802 Dosing Regimen Z

SUMMARY:
The purpose of this study is to assess the antiviral activity of JNJ-64281802 versus placebo in terms of reduction of dengue virus 1 (DENV-1) ribonucleic acid (RNA) viral load (VL).

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history, and vital signs performed at screening. If there are abnormalities, the participant may be included only if the investigator judges the abnormalities to be not clinically relevant. This determination must be recorded in the participant's source documents and initialed and dated by the investigator
* Must pass the comprehension test (i.e., obtain a passing score of greater than or equal to (>=) 75 percent (%), with up to 3 attempts in total) indicating that he or she understands the purpose, procedures, and potential risks and benefits of the study, after reading the informed consent and after the investigator or designee has provided detailed information on the study and answered the potential participant's questions
* Must have a blood pressure (after the participant is supine for >=5 minutes) between 90 and 140 millimeters of Mercury (mmHg) systolic, extremes included, and less than or equal to (<=) 90 mmHg diastolic at screening. Two repeat measurements are allowed in the absence of any other concerning health screening issues
* Must have a Body mass index (BMI) (weight in kilogram divided by the square of height in meters) between 18.0 and 33.0 kilogram per meter square (kg/m^2), extremes included, and a body weight of >=50.0 kg at screening
* All women of childbearing potential must have a negative highly sensitive serum (beta-human chorionic gonadotropin) pregnancy test at screening

Exclusion Criteria:

* Known allergies, hypersensitivity, or intolerance to JNJ-64281802 or its excipients, to a previous vaccination, or to specific medications/animals for which antigens may be in the dengue virus (DENV)-1 challenge strain preparations, including shellfish, fetal bovine serum, L-glutamine, neomycin, and streptomycin
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Received an investigational intervention (including investigational vaccines) or used an invasive investigational medical device within 6 months before first dose of study drug, or is currently enrolled in an investigational study, or is planning to be enrolled in an investigational study within 90 days after last dose of study drug
* Pregnant, breastfeeding, or planning to become pregnant during the study or within 90 days after last dose of study drug
* Plans to father a child during the study or within 90 days after last dose of study drug

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2027-09-02 (Estimated); Study Completion 2027-12-09 (Estimated)

PRIMARY OUTCOMES:
Area Under the DENV-1 RNA VL-concentration time Curve (VL AUC) from Immediately before Inoculation (Baseline on Day 1) until Day 29 | Baseline to Day 29
  Area under the dengue virus (DENV)-1 ribonucleic acid (RNA) Viral Load (VL) concentration-time curves from immediately before inoculation (baseline on Day 1) until Day 29 will be reported.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to Day 85
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with Clinically Significant Abnormalities in Physical Examination | Up to Day 85
  Number of participants with clinically significant abnormalities in physical examination will be reported.
Number of Participants with Clinically Significant Abnormalities in Vital Signs | Up to Day 85
  Number of participants with clinically significant abnormalities in vital signs (body temperature, pulse/heart rate, systolic and diastolic blood pressure) will be reported.
Number of Participants with Clinically Significant Abnormalities in Electrocardiogram (ECGs) | Up to Day 21
  Number of participants with clinically significant abnormalities in electrocardiogram (ECGs) will be reported.
Number of Participants with Clinically Significant Abnormalities in Laboratory Parameters | Up to Day 85
  Number of participants with clinically significant abnormalities in laboratory parameters (serum chemistry, hematology, blood coagulation, and urine samples) will be reported.
Number of Participants with DENV Infection Associated AEs | Up to Day 85
  Number of participants with DENV infection associated AEs will be reported.
Area Under the log10-transformed DENV 1 RNA VL Concentration-time Curves from Immediately before Inoculation (Baseline on Day 1) until Day 29 | Baseline to Day 29
  Area under the log10-transformed DENV 1 RNA VL concentration-time curves from immediately before inoculation (baseline on Day 1) until Day 29 will be reported.
Peak of Detectable DENV-1 RNA | Up to Day 85
  Peak of detectable DENV-1 RNA will be reported.
Duration of Detectable DENV-1 RNA | Up to Day 85
  Duration of detectable DENV-1 RNA will be reported.
Time to First Onset of Detectable DENV-1 RNA | Up to Day 85
  Time to first onset of detectable DENV-1 RNA will be reported.
Number of Participants with Detectable DENV-1 RNA | Up to Day 85
  Number of participants with detectable DENV-1 RNA will be reported.
Area Under the Viremia Curves from Immediately before Inoculation (Baseline on Day 1) until Day 29 | Baseline to Day 29
  Area under the viremia curves from immediately before inoculation (baseline on Day 1) until Day 29 will be reported.
Area Under the log10-transformed Viremia Curves | Up to Day 85
  Area under the log10-transformed viremia curves will be reported.
Peak of Detectable Viremia Level | Up to Day 85
  Peak of detectable viremia level will be reported.
Duration of Detectable Viremia | Up to Day 85
  Duration of detectable viremia will be reported.
Time to First Onset of Detectable Viremia | Up to Day 85
  Time to first onset of detectable viremia will be reported.
Number of Participants with Detectable Viremia | Up to Day 85
  Number of participants with detectable viremia will be reported.
Maximum Observed Analyte Concentration (Cmax) of JNJ-64281802 | Day -5: Predose, 1, 2, 4, 6, 8, 10, 12 hours Postdose; Day 21: Predose, 1, 2, 4, 6, 8, 12, 24 and 96 hours Postdose
  Cmax is the maximum observed analyte concentration.
Minimum Observed Analyte Concentration (Cmin) of JNJ-64281802 | Day 21: Predose, 1, 2, 4, 6, 8, 12, 24 and 96 hours Postdose
  Cmin is the minimum observed analyte concentration.
Trough Plasma Analyte Concentration (Ctrough) of JNJ-64281802 | Day -4, 1, 6, 8, 10, and 15: Predose; Day 21: Predose, 1, 2, 4, 6, 8, 12, 24 and 96 hours Postdose
  (Ctrough) is defined as observed analyte concentration just prior to the beginning or at the end of a dosing interval.
Average Analyte Concentration (Cavg) of JNJ-64281802 | Day -5: Predose, 1, 2, 4, 6, 8, 10, 12 hours postdose; Day 21: Predose, 1, 2, 4, 6, 8, 12, 24 and 96 hours Postdose
  Cavg is defined as average analyte concentration over the dosing interval (tau) and will be calculated as AUCtau/Tau.
Time to Reach Maximum Observed Plasma Analyte Concentration (Tmax) of JNJ-64281802 | Day -5: Predose, 1, 2, 4, 6, 8, 10, 12 hours postdose; Day 21: Predose, 1, 2, 4, 6, 8, 12, 24 and 96 hours Postdose
  Tmax is defined as the actual sampling time to reach the maximum observed plasma analyte concentration.
Fluctuation Index (FI) of JNJ-64281802 | Day 21: Predose, 1, 2, 4, 6, 8, 12, 24 and 96 hours Postdose
  FI is the percentage fluctuation (variation between maximum and minimum concentration at steady state), calculated as: 100*([Cmax-Cmin]/Cavg).
Area Under the Curve from Time Zero to End of Dosing Interval (AUCtau) | Day -5: Predose, 1, 2, 4, 6, 8, 10, 12 hours postdose; Day 21: Predose, 1, 2, 4, 6, 8, 12, 24 and 96 hours Postdose
  The AUCtau is the measure of the plasma analyte concentration from time zero to end of dosing interval. AUC during a dosing interval (τ), calculated by linear-linear trapezoidal summation.
Number of Participants with Anti DENV-1 Total IgM and IgG Antibody Titers | Up to Day 85
  Anti-DENV-1 immunoglobulin G (IgG) and immunoglobulin M (IgM) antibodies will be measured using enzyme-linked immunosorbent assay (ELISA).
Time to First Onset of Anti-DENV-1 Total IgM and IgG Antibody Titers | Up to Day 85
  Time to first onset of anti-DENV-1 total IgM and IgG antibody titers will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency